CLINICAL TRIAL: NCT06539325
Title: Rapid Molecular Diagnosis and Detection of Emerging Infectious Diseases in Patients With Tropical Fever
Brief Title: Rapid Molecular Diagnosis and Detection of Emerging Infectious Diseases in Patients With Tropical Fever (Tropifever)
Acronym: Tropifever
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: APHP231161
Record Dates: First submitted 2024-07-11; First posted 2024-08-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2024-08

CONDITIONS: Infectious Diseases in Febrile Patients Returning From Tropical Countries
Keywords: Tropical fever; Respiratory viruses; Arboviruses; Emerging infectious disease
MeSH Terms: conditions — Communicable Diseases, Emerging

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention period (Experimental): Patient management will be guided by a systematic microbiological diagnostic strategy
  Interventions: Diagnostic Test: Diagnosis algorithm according to the delay between travel and consultation
- Control period (No Intervention): Patient management will be done according to the usual practices of centers and emergency physicians

INTERVENTIONS:
Diagnostic Test: Diagnosis algorithm according to the delay between travel and consultation — Tests : RT-PCR for the most common arboviruses (Dengue, Zika, Chikungunya, and West Nile virus) and serology for dengue infection (NS1 antigen, and IgM and IgG), serologies for chronic viral infections (HIV, HBV and HCV) and schistosomiasis, Blood cultures and Innovativ Diagnostics : panel Dragonfly and two metagenomic analyses
  Arms: Intervention period

SUMMARY:
Travellers returning from tropical countries often present to emergency departments with acute fever. While systematic screening for malaria is well established in clinical practice in France, further diagnostic testing for infectious diseases is less codified. In addition, the clinical presentation of many tropical and emerging infectious diseases is often similar, making a positive diagnosis in these patients challenging.

Improving the microbiological diagnostic strategy for febrile travellers is crucial because the lack of an accurate diagnosis in many of these patients prevents the implementation of appropriate diagnostic and therapeutic measures. These measures include antimicrobial treatment, but also additional investigations, specialised monitoring and the initiation of follow-up of acute or chronic infections.

In addition, the current diagnostic approach to tropical fevers is poorly suited to detect outbreaks associated with a new or re-emerging infectious disease and to alert public health authorities in a timely manner.

Therefore, this project aims to evaluate the impact of a systematic and expanded microbiological diagnostic strategy for patients presenting to the emergency department with fever after returning from tropical countries. To evaluate this testing strategy, the investigators propose to conduct a multicentre, cluster-randomised, cross-over trial comparing standard care with a systematic microbiological diagnostic algorithm added to standard care.

DETAILED DESCRIPTION:
Frequently, travelers returning from tropical countries seek medical advice in the emergency department (ED) for acute fever. While the systematic search for malaria is well anchored in clinical practice in France, further diagnostic testing for infectious diseases (ID) is less codified. Besides, the clinical presentation of many tropical and emerging infectious pathologies (EID) is often similar, presenting challenges for a positive diagnosis in those patients.

Indeed, besides testing for malaria all patients with fever and a travel history in tropical regions in the last 3 months, there are, to our knowledge, no French guidelines on the diagnosis strategy of fever in the returning traveler. A few studies have proposed a syndromic testing strategy for patients admitted to ICU, but literature still lacks data on the efficiency of syndromic testing strategies in patients without severity criteria consulting at the ED. Other expert committees and literature on the topic usually recommend to collect a detailed clinical history including nature of travel, relevant activities and exposure, and physical findings, and then prescribe laboratory tests according to each situation. However, this common-sense clinical approach may not be adapted to the peculiar situation of emergency departments where the expertise of clinicians in infectious and tropical diseases may vary and time constraints do not always allow clinicians to collect a detailed history and examination. Moreover, even a careful medical history and physical examination may mislead clinicians in case of atypical clinical presentations or unexpected infections.

A recent study conducted in Spain, Switzerland and Belgium has shown that among travelers with acute undifferentiated febrile illnesses, 132/455 (29.0%) had viral infections, including 108/455 (23.7%) arboviruses, 96/455 (21.1%) malaria and 82/455 (18.0%) bacterial infections. A review of travel-related infections in 103,739 patients consulting in different European clinics between 1998 and 2018 reported an increase in arboviral infections over the last decade, with dengue, chikungunya and zika virus infections being almost as frequent as malaria between 2013 and 2018. A similar percentage of patients presented a viral syndrome with or without rash, in which the etiological agent could not be identified, emphasizing the gaps in our current testing strategy.

The diagnosis of respiratory viruses, including SARS-CoV-2, influenza, and respiratory syncytial virus (RSV), is often overlooked in returning travelers consulting in the emergency department (ED), despite being transmitted either year-long in tropical countries or during the rainy season, concomitantly with malaria. Rickettsial diseases, such as spotted fever or scrub typhus for example, represented 2% of febrile returning travelers in a recent article but are exceptionally sought after in the diagnostic process of patients consulting in the emergency department. Some of these patients with rickettsial diseases had no characteristic eschar. Likewise hemorrhagic fevers and, particularly Lassa fever, whose prevalence has been increasing in recent years in Nigeria are seldomly tested.

It is thus an open question whether a broader and more systematic microbiological laboratory testing strategy could enhance the number of diagnosis and thus the management of patients in this population. Indeed, improving our diagnostic strategy is crucial because the lack of a precise diagnosis in many of these patients prevents the implementation of appropriate diagnostic therapeutic measures. These measures obviously include antimicrobial treatments, but also additional investigations, specialized monitoring, and the initiation of a follow-up of acute or chronic infections. Indeed, the visit in the ED of those febrile travelers represents a unique opportunity to screen for chronic viral infections (such as HIV, hepatitis B and C), as well as acute hepatitis due to HAV or HEV, as this population of travelers is particularly at risk.

Potential measures also include isolation measures or public health measures such as mandatory reporting. Indeed, even though epidemiological surveillance systems and mandatory reporting have been established for dengue fever, chikungunya and other arboviruses, the number of reported cases in metropolitan France remains low and is probably underestimated. This limited testing in returning travelers impairs our ability to detect cryptic transmission of these diseases. Even though most of those infections are self-limiting, improving the detection of these arboviral infections is crucial, as their vectors, notably Aedes albopictus, are now present seasonally or yearlong in different French metropolitan areas. Thus, infected patients could potentially fuel local transmissions of arboviruses, emphasizing the need for improved diagnostic tools in metropolitan hospitals.

Furthermore, the current diagnosis approach for tropical fever is poorly suited to detect outbreaks linked to a new or re-emerging infectious disease and to promptly alert public health authorities. Although the diagnostic of viral hemorrhagic fevers for example is unlikely in returning travelers, the current diagnosis approach does not permit the early diagnosis of an outbreak, especially in the case of a pauci-symptomatic patient. Other emerging infectious diseases, such as shown by the recent example of Monkeypox, are never routinely screened before an outbreak occurs. However, recent data suggest that Monkeypox may have been circulating at low levels in France before the alert was given.

This project thus aims to evaluate the clinical impact of a systematic diagnostic strategy for patients consulting the ED for fever after returning from the tropics. To evaluate this testing strategy, the investigators propose to perform a multicentric, cluster-randomized trial comparing the standard of care with a systematic microbiological diagnostic algorithm added to the standard of care.

As discussed above, there is no well-established standard of care nor guidelines for the diagnostic approach of a returning traveler with fever in the emergency department. Literature exist but mostly consist of expert advice. Indeed, fever in a returning traveler is a complex condition with multiple potential diagnoses. The diagnostic approach in the emergency department is individualized, very heterogeneous and often limited by time constraints.

This is why the design proposed is a cluster randomized trial comparing Standard of Care (SoC) to Standard of Care plus a systematic microbiological diagnostic algorithm.

During intervention periods, this algorithm will be added to the SoC for every traveler returning from tropical countries and presenting with fever measured at the ED.

The investigators make the hypotheses that this project will:

1. improve the diagnosis of tropical and emerging infectious diseases in patients with a fever returning from tropical countries by using a systematic microbiological diagnostic approach
2. by providing microbiologically confirmed diagnosis, optimize the clinical management of patients including but not limited to additional investigations, specific monitoring, dedicated follow-up, isolation measures, antimicrobial treatment, thus improving patients' clinical outcomes
3. increase the application of public health measures for infectious and tropical diseases including mandatory reporting to the Regional Health Agency, thus improving the national surveillance of selected diseases
4. provide the participating centers with tools for the early detection of emerging infectious diseases, allowing them to participate in the surveillance and early alert of any emergence. Indeed, this protocol, by using and evaluating innovative and versatile diagnostic tools, is adapted to the rapid addition of one or multiple additional pair of primers into the diagnosis strategy in case of a new emergence or a re-emerging infectious disease.

Finally, the proposed microbiological diagnostic strategy and the precise analysis of microbiologically confirmed positive diagnosis in this study may inform future guidelines for the screening of infectious and tropical diseases in febrile returning travellers.

The investigators plan to include patients consulting in the emergency department for fever within 28 days of returning from tropical regions who do not have sepsis (qSOFA < 2) nor require immediate hospitalization.

Patients will be included in the emergency department because they usually are less explored than in other contexts such as a dedicated ID consultation. Moreover, studies have shown that patients seeking the ED are usually more frail or vulnerable than other patients. They visit the ED because they are often unaware of consultations dedicated to tropical pathologies and sometimes because they do not have a general practitioner. So the ED visit represents an excellent opportunity to put these patients back into an appropriate care plan. Patients will not be included in other contexts such as the outpatient clinic of infectious diseases because the standard of care in these structures might be different from emergency departments.

* Fever will be defined as a tympanic temperature above 38°c measured in the emergency department.
* The 28 days cut-off is based on the fact that most arboviruses, respiratory viruses and hemorrhagic fevers have a combined incubation and detection period below 28 days.
* Tropical regions will be defined as any region located between the Tropic of Cancer and the Tropic of Capricorn.
* Patients with sepsis (qSOFA ≥ 2) or patients who require hospitalization will not be included because they usually have rapid access to a wide panel of diagnostic testing while hospitalized and are explored more than patients who do not require hospitalization. Quick SOFA is widely used as a score for sepsis.

Standard of care is the standard diagnostic approach for returning travelers with fever. It will include the standard clinical evaluation of a patient with the collection of medical history, travel history, physical examination, etc. In addition to travel-related infections, cosmopolitan causes of fever should be considered in ill travellers, as well as non-infectious cause of fever including e.g. venous thrombosis, allergic fever, cancer, etc. The standard of care for diagnosis in a patient with fever is thus complex and heterogeneous among patients.

Regarding laboratory work-up, there are no specific guidelines for these patients, apart from systematic malaria testing. Standard of care usually includes systematic malaria thin smear +/- antigen test +/- qPCR, according to each center and local capacities sample for upper respiratory tract symptoms, chest X-Ray for abnormal auscultation, etc.

As part of this study, all patients included in the control period and the intervention period will have a follow-up visit planned with an infectious diseases' specialist at Day 4 +/-1.

The follow-up visit will allow clinicians to provide a diagnosis to the patient if a diagnosis has been confirmed and to organize subsequent diagnosis and therapeutic management of the patients. Day 4 +/-1 has been chosen for the follow-up visit because this ensures that the ID specialist will have access to most of the microbiological examinations included in the diagnostic algorithm, both in the control and in the intervention periods, and complies with the recommendation to see all patients with a diagnosis of malaria for the Day 3 monitoring.

The testing strategy that will be evaluated during this study includes tests that will be realized in all centres, in order to be available during the follow-up consultation with the ID specialist, and specialized tests that will be performed retrospectively in one central hospital (Bichat-Claude Bernard).

ELIGIBILITY:
Inclusion Criteria:

* Adult (age ≥ 18 years old)
* Fever (tympanic temperature above 38°c measured in the emergency department)
* Within 28 days of returning from tropical countries (Sub-Saharan Africa, South and Southeast Asia, Central and South America)
* No sepsis (qSOFA < 2)

Exclusion Criteria:

* Patient requiring hospitalization
* Patient unable to consent: unconscious or language barrier without an available translator
* Patient under legal protection measure (guardianship, curatorship, legal protection, deprivation of liberty, hospitalisation for psychiatric care)
* Patient refusing to participate

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 564 (Estimated)
Dates: Start 2024-08-26 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of Patient informed of a microbiologically confirmed infection and of the appropriate course of action within five days after the initial visit to the emergency department. | 5 days
  Number of Patient informed of a microbiologically confirmed infection and of the appropriate course of action within five days after the initial visit to the emergency department.

SECONDARY OUTCOMES:
Number of Patient with a microbiologically confirmed diagnosis within 5 days after ED visit. | 5days
  Number of Patient with a microbiologically confirmed diagnosis within 5 days after ED visit.
Number of Lost to follow up patient: a patient will be considered lost to follow up if no contact has been established to informed him of the result of the diagnostic tests within 5 days after ED visit (neither by phone nor during a hospital visit). | 3 months
  Number of Lost to follow up patient: a patient will be considered lost to follow up if no contact has been established to informed him of the result of the diagnostic tests within 5 days after ED visit (neither by phone nor during a hospital visit).
Number of Hospitalizations linked to the diagnosis, according to the physician in charge, in the 3 months following inclusion | 3 months
  Number of Hospitalizations linked to the diagnosis, according to the physician in charge, in the 3 months following inclusion
Mortality at 3 months following ED visit, mortality linked to the diagnosis according to the investigator or the physician in charge of the patient at 3 months following ED visit | 3 months
  Mortality at 3 months following ED visit, mortality linked to the diagnosis according to the investigator or the physician in charge of the patient at 3 months following ED visit
Number of the specific management of patients | 3 months
  including:
  * Additional investigations
  * Systematic monitoring (e.g., thrombocytopenia in case of dengue fever)
  * Dedicated long-term follow-up (e.g., HIV follow-up)
  * Antimicrobial treatments
  * Isolation measures
  * Family screening
  * Public health measures such as mandatory reporting (signalling and notification)
Total Cost of the strategy of infectious disease management | 3 months
  Total Cost of the strategy of infectious disease management
Diagnostic performances of the Dragonfly panel compared to reference PCR panel: sensitivity, specificity, positive and negative predictive values will be calculated | 3 months
  Diagnostic performances of the Dragonfly panel compared to reference PCR panel: sensitivity, specificity, positive and negative predictive values will be calculated
Delay (number of days) in the addition of a new set of primers in the Dragonfly panel | 3 months
  In the case of the emergence of a new respiratory pathogen, such as SARS-CoV-2 in 2019, additional secondary endpoints will be added
Diagnostic performance of the new set of primers integrated into the Dragonfly panel compared to the PCR developed by the French and international reference centers (sensitivity, specificity, positive predictive value, negative predictive value) | 3 months
  In the case of the emergence of a new respiratory pathogen, such as SARS-CoV-2 in 2019, additional secondary endpoints will be added
Length of hospitalizations linked to the diagnosis, according to the physician in charge, in the 3 months following inclusion | 3 months
  Length of hospitalizations linked to the diagnosis, according to the physician in charge, in the 3 months following inclusion
Total cost of compliance with the diagnostic workup | 3 months
  Total cost of compliance with the diagnostic workup
Number of hospitalizations and linked mortality at 3months | 3 months
  Number of hospitalizations and linked mortality
Number of death at 3 months | 3 months
  Number of death at 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Service des Urgences, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No